CLINICAL TRIAL: NCT06360731
Title: The Effect of 4-7-8 Breathing Exercise Technique on Tinnitus Handicap, Psychological Factors, and Sleep Quality in Tinnitus Patients: A Randomized Controlled Study
Brief Title: The Effect of 4-7-8 Breathing Exercise Technique on Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gulce Kirazli, Asst.Prof., Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1018
Record Dates: First submitted 2024-04-05; First posted 2024-04-11 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Tinnitus, Subjective
Keywords: 4-7-8 breathing exercise; Tinnitus; Psychological factors; Insomnia; Informative session
MeSH Terms: conditions — Tinnitus; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This study employs a parallel group randomised controlled trial design.
Who Masked: Participant, Investigator
Masking Description: In the study, patients do not know which group they were in. Therefore, blinding is performed among the participants. To prevent bias in the study, blinding is also performed between the researchers. Researchers (S.B. and A.O. from both clinics) make the pre- and post-test evaluations without knowing which group the patients are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Experimental group who consists of subjective tinnitus patients will receive 1 hour of informative session on tinnitus and also perform 4-7-8 breathing exercises for 6 weeks
  Interventions: Other: 4-7-8 breathing exercise technique and informative session on tinnitus
- Control Group (Active Comparator): Control group who consists of subjective tinnitus patients will receive 1 hour of informative session on tinnitus only
  Interventions: Other: Informative session on tinnitus

INTERVENTIONS:
Other: 4-7-8 breathing exercise technique and informative session on tinnitus — Participants in experimental group will be individually provided with informative session on tinnitus for one hour by researchers. During the informative session, the participants will be given general information about tinnitus and will be informed about the possible causes, symptoms, diagnosis, therapy, or treatment processes, and coping methods. The participants will be also given a printed informative brochure on tinnitus. In the same session, after one hour of informative session, the 4-7-8 breathing exercise method will be demonstrated by the same researchers. In addition, a video showing how to perform the 4-7-8 breathing exercise technique will be sent as a text message to their cell phones.
  Arms: Experimental Group
Other: Informative session on tinnitus — Participants in control group will be individually provided with informative session on tinnitus only for one hour by researchers G.K. and G.S.U. from both clinics. During the informative session, the participants will be given general information about tinnitus and inform about the possible causes, symptoms, diagnosis, therapy, or treatment processes, and coping methods. The participants will be also given a printed informative brochure on tinnitus.
  Arms: Control Group

SUMMARY:
The goal of this study is to evaluate the effect of 4-7-8 breathing exercise on tinnitus handicap, psychological factors and sleep quality.

There will be a parallel-group randomized controlled trial study and consists of two groups.

Both groups will receive 1 hour of informative session on tinnitus and the experimental group will also perform 4-7-8 breathing exercises for 6 weeks. Visual analog scale, tinnitus handicap inventory, insomnia severity index, trait anxiety inventory, and perceived stress scale will be applied before and after the application.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of 4-7-8 breathing exercise technique on tinnitus handicap, psychological factors and sleep quality. It is also aimed to compare the results of the experimental group and those who received only 1 hour of informative session on tinnitus (Control group).

The study will employ a parallel-group randomized controlled trial design. Both groups will receive 1 hour of informative session on tinnitus and the experimental group will also perform 4-7-8 breathing exercises for 6 weeks.

Visual analog scale, tinnitus handicap inventory, insomnia severity index, trait anxiety inventory,and perceived stress scale will be applied to all patients before and after the application.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65 years with subjective idiopathic tinnitus complaints for at least six months
* Must be able to speak and read Turkish
* Must be able to answer the questionnaire questions and perform the 4-7-8 breathing exercises regularly

Exclusion Criteria:

* Any neuro-otologic, psychiatric, neurologic, or cognitive problems, objective tinnitus, chronic medication use, asthma diagnosis or respiratory distress
* Receivement of any tinnitus treatment or tinnitus informative session actively

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline
  Patients will be asked to assess the degree of distress and annoyance associated with their tinnitus, as well as its severity, using a Visual Analog Scale (VAS) from 0 to 10 both before and after the application. An increase in these areas is shown by an increase in the score. Minimum score value is 0 and maximum value is 10. All patients will be assessed before application.
Visual Analog Scale (VAS) | Six weeks after baseline evaluation
  Patients will be asked to assess the degree of distress and annoyance associated with their tinnitus, as well as its severity, using a Visual Analog Scale (VAS) from 0 to 10 both before and after the application. An increase in these areas is shown by an increase in the score. Minimum score value is 0 and maximum value is 10. All patients will be assessed six weeks after baseline evaluation.
Tinnitus Handicap Inventory (THI) | Baseline
  The Tinnitus Handicap Inventory (THI) assesses the catastrophic, emotional, and functional impacts of tinnitus and measures its effects on patients' daily functioning. The THI consists of 25 items. In the inventory, there are 25 items consisting of three options as 'yes', 'no', and 'sometimes'. A 'yes' answer is worth 4 points and a 'no' answer is worth 0 points. A maximum score of 100 points can be obtained from the THI. The higher the score, the greater the perception of the tinnitus as a handicap. Minimum score value is 0 and maximum value is 100. All patients will be assessed before application.
Tinnitus Handicap Inventory (THI) | Six weeks after baseline evaluation
  The Tinnitus Handicap Inventory (THI) assesses the catastrophic, emotional, and functional impacts of tinnitus and measures its effects on patients' daily functioning. The THI consists of 25 items. In the inventory, there are 25 items consisting of three options as 'yes', 'no', and 'sometimes'. A 'yes' answer is worth 4 points and a 'no' answer is worth 0 points. A maximum score of 100 points can be obtained from the THI. The higher the score, the greater the perception of the tinnitus as a handicap. Minimum score value is 0 and maximum value is 100. All patients will be assessed six weeks after baseline evaluation.
Insomnia severity index (ISI) | Baseline
  Sleep quality of the patients was assessed with the insomnia severity index (ISI). It is a questionnaire that evaluates the difficulties experienced in transitioning to and maintaining sleep, the level of stress caused by sleep problems, and impairments in daily functions, and thus determines the level of insomnia. It consists of 7 questions in total. Higher score indicates more insomnia symptoms. Minimum score value is 0 and maximum value is 28. All patients will be assessed before application.
Insomnia severity index (ISI) | Six weeks after baseline evaluation
  Sleep quality of the patients was assessed with the insomnia severity index (ISI). It is a questionnaire that evaluates the difficulties experienced in transitioning to and maintaining sleep, the level of stress caused by sleep problems, and impairments in daily functions, and thus determines the level of insomnia. It consists of 7 questions in total. Higher score indicates more insomnia symptoms. Minimum score value is 0 and maximum value is 28. All patients will be assessed six weeks after baseline evaluation.
Perceived stress scale -10 (PSS-10) | Baseline
  The Perceived Stress Scale-10 (PSS-10) will be administered to assess the stress perceived by tinnitus patients. It was developed to measure the extent to which situations in one's life are considered stressful. It consists of 10 questions. The scores of PSS-10 vary between 0 and 40. Greater perceived stress is indicated by higher scores. The scores of PSS-10 vary between 0 and 40. All patients will be assessed before application.
Perceived stress scale -10 (PSS-10) | Six weeks after baseline evaluation
  The Perceived Stress Scale-10 (PSS-10) will be administered to assess the stress perceived by tinnitus patients. It was developed to measure the extent to which situations in one's life are considered stressful. It consists of 10 questions. The scores of PSS-10 vary between 0 and 40. Greater perceived stress is indicated by higher scores. The scores of PSS-10 vary between 0 and 40. All patients will be assessed six weeks after baseline evaluation.
Trait Anxiety Scale (TAS) | Baseline
  The trait anxiety subscale of the State-Trait Anxiety Inventory was used to assess the level of anxiety in those with tinnitus. The TAS is a 4-point Likert-type scale consisting of twenty items that aims to determine how the individual feels regardless of the situation and conditions in which they find themselves. A score between 20 and 80 is obtained from this scale. Higher scores indicate higher level of anxiety. A score between 20 and 80 is obtained from this scale. All patients will be assessed before application.
Trait Anxiety Scale (TAS) | Six weeks after baseline evaluation
  The trait anxiety subscale of the State-Trait Anxiety Inventory was used to assess the level of anxiety in those with tinnitus. The TAS is a 4-point Likert-type scale consisting of twenty items that aims to determine how the individual feels regardless of the situation and conditions in which they find themselves. A score between 20 and 80 is obtained from this scale. Higher scores indicate higher level of anxiety. A score between 20 and 80 is obtained from this scale. All patients will be assessed six weeks after baseline evaluation.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Gokce Saygi Uysal, Ankara
  - Audiology Unit of the Department of Otorhinolaryngology, Ege University Faculty of Medicine Hospital, Izmir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koksoy S, Eti CM, Karatas M, Vayisoglu Y. The Effects of Yoga in Patients Suffering from Subjective Tinnitus. Int Arch Otorhinolaryngol. 2018 Jan;22(1):9-13. doi: 10.1055/s-0037-1601415. Epub 2017 Apr 3. PMID 29379573
- [Background] Vierra J, Boonla O, Prasertsri P. Effects of sleep deprivation and 4-7-8 breathing control on heart rate variability, blood pressure, blood glucose, and endothelial function in healthy young adults. Physiol Rep. 2022 Jul;10(13):e15389. doi: 10.14814/phy2.15389. PMID 35822447
- [Result] Gilles A, Jacquemin L, Cardon E, Vanderveken OM, Joossen I, Vermeersch H, Vanhecke S, Van den Brande K, Michiels S, Van de Heyning P, Van Rompaey V. Long-term effects of a single psycho-educational session in chronic tinnitus patients. Eur Arch Otorhinolaryngol. 2022 Jul;279(7):3301-3307. doi: 10.1007/s00405-021-07026-7. Epub 2021 Oct 1. PMID 34596715
- [Result] Apoorva HM, Jayaram M, Patil NJ. Usefulness of Yoga in the management of tinnitus during COVID-19: A narrative review. J Ayurveda Integr Med. 2024 Jan-Feb;15(1):100822. doi: 10.1016/j.jaim.2023.100822. Epub 2023 Dec 28. PMID 38157657
- [Result] Ismail AMA, Ali SM, Ghuiba K, Elfahl AMA, Tolba AMN, Ghaleb HAM. Autonomic functions, tinnitus annoyance and loudness, and quality of life: Randomized-controlled responses to bee-humming (vibrational) respiratory training in tinnitus elderly. Complement Ther Clin Pract. 2022 Aug;48:101611. doi: 10.1016/j.ctcp.2022.101611. Epub 2022 Jun 3. PMID 35675742
- [Result] Gunjawate DR, Ravi R. Effect of yoga and meditation on tinnitus: a systematic review. J Laryngol Otol. 2021 Apr;135(4):284-287. doi: 10.1017/S0022215121000566. Epub 2021 Mar 11. PMID 33691808
- [Result] Video: breathing exercises: 4-7-8 breath [Internet]. 2014 Available from: https://www.drweil.com/videos-features/videos/breathing-exercises-4-7-8-breath/
- [Result] Aksoy S, Firat Y, Alpar R. The Tinnitus Handicap Inventory: a study of validity and reliability. Int Tinnitus J. 2007;13(2):94-8. PMID 18229787
- [Result] Boysan M, Güleç M, Beşiroğlu L, et al. Psychometric properties of the Insomnia Severity Index in Turkish sample. Anadolu Psikiyatri Derg 2010;11:248-252.
- [Result] Eskin M, Harlak H, Demirkıran F. The adaptation of the perceived stress scale into turkish: a reliability and validity analysis. Neuropsych Investig 2013;51:132-140.
- [Result] Öner N, Lecompte A. Manual of state trait anxiety inventory. Istanbul: Boğaziçi University Print House; 1998.